CLINICAL TRIAL: NCT01523210
Title: Influence of Physiotherapy on the Spastic Musculus Biceps Brachii Under Routine Botulinum Toxin Injection. - An Explorative MRI Study
Brief Title: DTI Study of the Influence of Physiotherapy on Distribution of BoNT in Spastic Muscle
Status: Completed | Type: Observational
Sponsor: Kirsten Elwischger, MD (Other)
Responsible Party: Sponsor-Investigator, Kirsten Elwischger, MD, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: DTI_BoNT_distribution
Record Dates: First submitted 2012-01-07; First posted 2012-02-01 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Spasticity
Keywords: spasticity; Diffusor tensor imaging; distribution; botulinum toxin; physiotherapy
MeSH Terms: conditions — Muscle Spasticity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- upper limb spasticity: patients suffering from upper limb spasticity and are treated with botulinum toxin
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — thirty minutes passive flexion and extension of the elbow joint by a physiotherapist
  Other Names: physical therapy

SUMMARY:
Intramuscular application of botulinum toxin (BoNT) is used as a successful therapy of muscle spasticity. Clinical practice shows, that even with the use of special guidance techniques to increase accuracy of targeting, BoNT may spread to adjacent sites by diffusion. This causes fluctuating treatment response, unintended side effects, and decrease of effect due to production of antibodies. Hence, clinicians require increase of efficacy and safety by dose reduction, improvement of injection technique, and additional treatment strategies. Referring to this, animal model showed increased efficacy and decreased systemic side effects of BoNT in the injected muscle after active or passive manipulation of muscle. The mechanism of this effect remain unclear.

T2 and (Diffusion Tensor Imaging) DTI technique can evaluate the in-vivo distribution of fluids in human skeletal muscle. In addition, it allows to differentiate denervated muscle tissue, caused by BoNT injections, from surrounding unaffected muscle tissue.

Up to the investigators knowledge, neither a human, in vivo measurement of the influence of passive muscle activity on the area of denervation, nor the primary, in-vivo distribution of BoNT within spastic human muscle tissue, been evaluated.

The aim of this explorative study is:

* to monitor the inflow and regional distribution of the injection bolus by dynamic T2-weighted-, DTI-sequences;
* to assess the effect of passive muscle exercise on the area of denervated, caused by BoNT, measured by DTI-, T2-weighted and flair sequences.

The investigators hypothesize, that

* intramuscular denervation area, measured by DTI-, T2-weighted and Fluid Attenuated Inversion Recovery (FLAIR) sequences, 3 weeks after routine BoNT injection, is facilitated by passive muscle exercise;
* primary distribution of the injected BoNT bolus can be non-invasively monitored by dynamic T2-, DTI- and T2 weighted sequences.

Therefore, in this investigator blinded, cross-over study, 6 patients suffering from upper limb spasticity, including musculus biceps brachii, will be investigated. (Magnetic Resonance Tomography) MRI of the musculus biceps brachii will be performed at two consecutive, routine BoNT-injection days (baseline and week 16). Patients receive dosage as clinically indicated, due to routine treatment. Patients will be randomised to receive thirty minutes of physiotherapy of the affected arm, including exercise of the elbow flexors, at one of the injection days (baseline, or week 16, respectively). In addition, MRI will be repeated 3 weeks after injection.

DETAILED DESCRIPTION:
* At baseline and week 16, dynamic T2-, T2-,and DTI weighted sequences will be performed to monitor the injection of the BoNT-bolus. Immediate after MRI-scan, physiotherapy will be performed. Patients, who were randomised to the non-treatment group at baseline, will receive physiotherapy immediately after MRI at week 16.
* At week 3 and week 19, three weeks after BoNT injection, respectively, MRI will be repeated. T2-and DTI- weighted and FLAIR- sequences will be performed.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in this clinical pilot trial
* age 18-80 years
* ≥4 months under routine botulinum toxin treatment
* last botulinum toxin treatment ≥3 months before screening
* spasticity of m. biceps brachii elbow flexion: Modified Ashworth Scale (MAS) ≥3

Exclusion Criteria:

* bleeding disorders or acute bleeding event.
* coumarine, warfarine therapy.
* non-MRI compatible medical (prothetics, pacemaker, etc) or non medical implantation (tattoos, intraorbital metal splinters, etc.) or other contraindications for MRI, not meeting the general safety recommendations for 3Tesla MRI.
* claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from upper limb spasticity
  receiving routine BoNT injection
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change of Fractionated Anisotropie (FA) value | baseline, week 3, week 16, week 19
  FA value reflects indirect diffusion
change of muscle cross-sectional area after routine botulinum toxin injection | baseline, week 3, week 16, week 19
  reflected by diameter of signal changes on T2-weighted and short-tau inversion recovery (STIR) sequences
Change of Apparent Diffusion Coefficient (ADC) values | baseline, week 3, week 16, week 19
  ADC describes structural changes of myocytes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sycha, Prof., MD, Principal Investigator — Medical University of Vienna, Department of Neurology
Locations (1):
- Medical University of Vienna, Department of Neurology, Vienna, Vienna, Austria